CLINICAL TRIAL: NCT07361380
Title: Non-Invasive Testing of Blood Biomarkers in Pregnant Women
Brief Title: Non-Invasive Testing Device for Anaemia
Acronym: NITA
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 24/WS/0122
Record Dates: First submitted 2026-01-13; First posted 2026-01-23 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy
Keywords: Pregnancy; Haemoglobin; Anaemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples will be analysed for a) whole blood, plasma and serum lipid and inflammatory marker analysis and b) iron studies and c) analysis of biochemistry and metabolism and d) analysis of biomarkers associated with inflammation, angiogenesis and endothelial, liver, and kidney function.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants who are pregnant.

SUMMARY:
Anaemia (iron deficiency) arises from a reduction in the number of healthy red blood cells or the level of haemoglobin (Hb) (a protein inside red blood cells) necessary to effectively transport oxygen throughout the body. Anaemia is common among pregnant women. The gold standard for anaemia diagnosis still relies on laboratory blood tests, which come with limitations in terms of point-of-care capability, accessibility and quality. The investigators have developed a portable and user-friendly device capable of detecting anaemia rapidly and non-invasively and facilitating appropriate treatment by distinguishing anaemia due to iron deficiency from other causes. The device, named The Vascular Imaging Tool for the Auricle (VITA), utilises high-resolution imaging technology to capture detailed images of blood cells and small blood vessels within the human body. The objectives of this study are to assess VITA's performance of (haemoglobin (Hb)) testing and its ability to identify iron deficiency anaemia against the clinical gold standard of laboratory blood tests.

DETAILED DESCRIPTION:
Anaemia arises from a reduction in the number of healthy red blood cells or the level of haemoglobin necessary to transport oxygen effectively throughout the body. It is a significant global health concern, affecting 1.6 billion individuals worldwide and untreated anaemia can contribute to chronic heart failure and chronic kidney disease. Anaemia is common among pregnant women. Mild cases of anaemia often go unnoticed due to their nonspecific symptoms, such as fatigue, headaches, and hair loss. Furthermore, studying this disease can be difficult as, particularly in places without ready access to laboratory blood sample analysis as current point-of-care solutions are not able to distinguish between different types of anaemia and prescribe suitable treatments. The gold standard for anaemia diagnosis still relies on laboratory blood tests, which come with limitations in terms of point-of-care capability, accessibility, and biases related to poor standardisation of assays and low sample quality.

The investigators have developed a portable and user-friendly device capable of detecting anaemia rapidly and non-invasively and facilitating appropriate treatment by distinguishing anaemia due to iron deficiency from other causes. The device, named The Vascular Imaging Tool for the Auricle (VITA), utilises high-resolution imaging technology to capture detailed images of blood cells and small vessels within the human body. Unlike existing non-invasive devices that can only measure properties in bulk tissue samples, VITA can analyse characteristics of hundreds of individual cells, thereby facilitating rapid point-of-care testing for iron deficiency anaemia. VITA is a low-cost device, and its unique ability to measure these parameters without requiring consumables or trained operators makes it particularly well-suited for researching anaemia in a range of settings, including low- and middle-income countries.

This project is a proof-of-concept study to assess VITA's performance of Hb testing. Secondary objectives include testing VITA's ability to identify iron deficiency anaemia against the clinical gold standard of laboratory blood tests, identification of other frequently measured blood biomarkers, and identification of biomarkers for long-term health. This study is not collecting data for licensing of the device.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Pregnant
* Aged 16-50 years

Exclusion Criteria:

* Ear piercings that cannot be temporarily removed that would prevent the ability of the VITA device to take images of the ear blood vessels.
* Ear piercings that would be visible on the ear blood vessel images

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Women who are pregnant
Study Population: Participants who are pregnant.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
To compare Hb measured by VITA with Hb measured by blood sample analysis | Baseline
  Agreement between the two measurements as calculated by systemic error (bias), and 95% limits of agreement as bias ±2 SD concentration of haemoglobin in the blood in g/dl of VITA and blood sample analysis

SECONDARY OUTCOMES:
To determine the maximum accuracy of VITA in detecting iron deficiency anaemia as compared to diagnosis based on guidelines on full iron studies in blood sample analysis | Baseline
  Accuracy of VITA algorithmic diagnosis (yes/no) compared to diagnosis (yes/no) based on haemoglobin, soluble transferrin receptor (sTfR), RDW (red cell distribution width), ferritin, serum iron, transferrin saturation (TSAT), mean corpuscular volume (MCV) and/or mean corpuscular haemoglobin concentration (MCHC)
To train image processing software to detect biomarkers that are frequently used in clinical practice based on VITA images | Baseline
  Correlation of VITA algorithmic metrics and blood sample analysis metrics of the following biomarkers:
  * Folate
  * Renal function
  * Electrolytes
  * Liver function
  * Calcium phosphate
  * Thyroid function
  * Full blood count
  * Glucose
  * Insulin
  * Lipids
  * HbA1C
To predict long-term health outcomes from features in VITA images | 6 months post-partum
  Medical records will be checked up to 6 months post-partum to check for the following indications:
  * Hypertensive disorders of pregnancy (gestational hypertension, pre-eclampsia, HELLP)
  * Other pregnancy complications
  * Blood pressure
  * Post-partum medical complications

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available